CLINICAL TRIAL: NCT02073656
Title: A Phase 3, Multicenter, Open-Label Study to Investigate the Efficacy and Safety of Sofosbuvir/Ledipasvir Fixed-Dose Combination for 12 Weeks in Subjects With Chronic Genotype 1 or 4 Hepatitis C Virus (HCV) and Human Immunodeficiency Virus (HIV)-1 Co-infection
Brief Title: Efficacy and Safety of Ledipasvir/Sofosbuvir Fixed-Dose Combination for 12 Weeks in Subjects With Chronic Genotype 1 or 4 HCV and HIV-1 Co-infection
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GS-US-337-0115
Record Dates: First submitted 2014-02-25; First posted 2014-02-27 (Estimated); Results first posted 2016-10-21 (Estimated); Last update posted 2018-11-16 (Actual); Status verified 2016-08

CONDITIONS: Hepatitis C Virus; HIV
Keywords: genotype 1; genotype 4; HIV
MeSH Terms: conditions — Hepatitis C | interventions — ledipasvir, sofosbuvir drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- LDV/SOF 12 Weeks (Experimental): LDV/SOF for 12 weeks
  Interventions: Drug: LDV/SOF
- Retreatment Substudy (Experimental): LDV/SOF plus RBV for 24 weeks
  Interventions: Drug: LDV/SOF; Drug: RBV

INTERVENTIONS:
Drug: LDV/SOF — 90/400 mg FDC tablet administered orally once daily
  Other Names: Harvoni®; GS-5885/GS-7977
Drug: RBV — Tablets administered orally in a divided daily dose according to package insert weight-based dosing recommendations (< 75 kg = 1000 mg and ≥ 75 kg = 1200 mg)
  Arms: Retreatment Substudy

SUMMARY:
This study will evaluate the antiviral efficacy, safety, and tolerability of ledipasvir/sofosbuvir (LDV/SOF) fixed-dose combination (FDC) administered for 12 weeks in hepatitis C virus (HCV) treatment-naive and treatment-experienced (including treatment intolerant) participants with chronic genotype 1 or 4 HCV infection who are co-infected with HIV-1.

Participants who experience confirmed post-treatment virologic failure (relapse) at or before Posttreatment Week 24 may be eligible to be enrolled in the Retreatment Substudy to receive LDV/SOF plus ribavirin (RBV) for 24 weeks.

ELIGIBILITY:
Inclusion Criteria:

* HCV RNA ≥ 10,000 IU/mL at screening
* HCV genotype 1 or 4
* HIV-1 infection
* Cirrhosis determination, a fibroscan or liver biopsy may be required
* Screening laboratory values within defined thresholds
* Use of protocol specified method(s) of contraception if female of childbearing potential or sexually active male

Exclusion Criteria:

* Clinically-significant illness (other than HCV or HIV) or any other major medical disorder that may interfere with subject treatment, assessment, or compliance with the protocol
* Current or prior history of clinical hepatic decompensation, hepatocellular carcinoma (HCC), or other malignancy (with the exception of certain resolved skin cancers)
* Hepatitis B virus (HBV) infection
* Pregnant or nursing female
* Chronic use of systemically administered immunosuppressive agents

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 335 (Actual)
Dates: Start 2014-02; Primary Completion 2014-11 (Actual); Study Completion 2015-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jenny Yang, PharmD, Study Director — Gilead Sciences
Locations (41):
- United States (34):
  - Birmingham, Alabama
  - Los Angeles, California
  - Newport Beach, California
  - Palo Alto, California
  - Sacramento, California
  - San Diego, California
  - San Francisco, California
  - Torrance, California
  - Denver, Colorado
  - Washington D.C., District of Columbia
  - Bradenton, Florida
  - Miami, Florida
  - Orlando, Florida
  - Tampa, Florida
  - Atlanta, Georgia
  - Decatur, Georgia
  - Chicago, Illinois
  - Lutherville, Maryland
  - Boston, Massachusetts
  - Kansas City, Missouri
  - Santa Fe, New Mexico
  - New York, New York
  - The Bronx, New York
  - Chapel Hill, North Carolina
  - Durham, North Carolina
  - Cincinnati, Ohio
  - Allentown, Pennsylvania
  - Philadelphia, Pennsylvania
  - Providence, Rhode Island
  - Dallas, Texas
  - Houston, Texas
  - Annandale, Virginia
  - Richmond, Virginia
  - Seattle, Washington
- Canada (4):
  - Vancouver, British Columbia
  - Ottawa, Ontario
  - Toronto, Ontario
  - Montreal, Quebec
- New Zealand (2):
  - Auckland
  - Christchurch
- San Juan, Puerto Rico

IPD SHARING:
Plan to Share IPD: Yes
Qualified external researchers may request IPD for this study after study completion. For more information, please visit our website at http://www.gilead.com/research/disclosure-and-transparency.
Supporting Information: Study Protocol, SAP
Time Frame: 18 months after study completion
Access Criteria: A secured external environment with username, password, and RSA code.
URL: http://www.gilead.com/research/disclosure-and-transparency

REFERENCES:
- [Result] Cooper C, Naggie S, Saag M, Yang JC, Stamm LM, Dvory-Sobol H, et al. Retreatment of Patients Who Failed 12 Weeks of Ledipasvir/Sofosbuvir-Based Regimens with Ledipasvir/Sofosbuvir with Ribavirin for 24 Weeks [Poster Presentation]. 23nd Conference on Retroviruses and Opportunistic Infections (CROI); 2016 February 22-25; Boston, MA.
- [Result] Naggie S, Cooper C, Saag M, Workowski K, Ruane P, Towner WJ, Marks K, Luetkemeyer A, Baden RP, Sax PE, Gane E, Santana-Bagur J, Stamm LM, Yang JC, German P, Dvory-Sobol H, Ni L, Pang PS, McHutchison JG, Stedman CA, Morales-Ramirez JO, Brau N, Jayaweera D, Colson AE, Tebas P, Wong DK, Dieterich D, Sulkowski M; ION-4 Investigators. Ledipasvir and Sofosbuvir for HCV in Patients Coinfected with HIV-1. N Engl J Med. 2015 Aug 20;373(8):705-13. doi: 10.1056/NEJMoa1501315. Epub 2015 Jul 21. PMID 26196665
- [Result] Naggie S, Cooper C, Saag M, Stamm LM, Yang JC, Pang PS, et al. Ledipasvir/Sofosbuvir for 12 Weeks in Patients Coinfected With HCV and HIV-1 [Oral Presentation]. 22nd Conference on Retroviruses and Opportunistic Infections (CROI); 2015 February 23-26; Seattle, WA.
- [Result] Cooper C, Naggie S, Saag M, Yang JC, Stamm LM, Dvory-Sobol H, Han L, Pang PS, McHutchison JG, Dieterich D, Sulkowski M. Successful Re-treatment of Hepatitis C Virus in Patients Coinfected With HIV Who Relapsed After 12 Weeks of Ledipasvir/Sofosbuvir. Clin Infect Dis. 2016 Aug 15;63(4):528-31. doi: 10.1093/cid/ciw349. Epub 2016 May 25. PMID 27225242
- [Derived] Saeed S, Strumpf EC, Walmsley SL, Rollet-Kurhajec K, Pick N, Martel-Laferriere V, Hull M, Gill MJ, Cox J, Cooper C, Klein MB; Canadian Co-Infection Cohort Study; Cohen J, Conway B, Cooper C, Cote P, Cox J, Gill J, Haider S, Harris M, Haase D, Hull M, Montaner J, Moodie E, Pick N, Rachlis A, Rouleau D, Sandre R, Tyndall JM, Vachon ML, Walmsley S, Wong D. How Generalizable Are the Results From Trials of Direct Antiviral Agents to People Coinfected With HIV/HCV in the Real World? Clin Infect Dis. 2016 Apr 1;62(7):919-926. doi: 10.1093/cid/civ1222. Epub 2016 Jan 6. PMID 26743093

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at study sites in the United States (including Puerto Rico), Canada, and New Zealand. The first participant was screened on 24 February 2014. The last study visit occurred on 01 December 2015.
Pre-assignment Details: 429 participants were screened.
Groups:
- LDV/SOF 12 Weeks: Ledipasvir/sofosbuvir (LDV/SOF) (90/400 mg) fixed-dose combination (FDC) tablet once daily for up to 12 weeks.
  Participants who experienced confirmed post-treatment virologic failure (relapse) at or before Posttreatment Week 24 were eligible to be enrolled in the Retreatment Substudy to receive LDV/SOF (90/400 mg) FDC tablet once daily + ribavirin (RBV) tablets (1000-1200 mg daily based on weight) for 24 weeks.
Period: Primary Study
Arm/Group | LDV/SOF 12 Weeks
Started | 335
Completed | 327
Not Completed | 8
Not completed — Lost to Follow-up | 6
Not completed — Death | 1
Not completed — Withdrew Consent | 1
Period: Retreatment Substudy
Arm/Group | LDV/SOF 12 Weeks
Started | 9 (Only participants experiencing virologic relapse in the Primary Study were eligible for retreatment.)
Completed | 9
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Safety Analysis Set: participants who enrolled and received at least 1 dose of study drug.
Groups:
- LDV/SOF 12 Weeks: Ledipasvir/sofosbuvir (LDV/SOF) (90/400 mg) fixed-dose combination (FDC) tablet once daily for up to 12 weeks.
Arm/Group | LDV/SOF 12 Weeks
Number analyzed (Participants) | 335
Age, Continuous [Mean (Standard Deviation); unit: years] | 52 (8.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 59
  Male | 276
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 56
  Not Hispanic or Latino | 276
  Unknown or Not Reported | 3
Race/Ethnicity, Customized [Number; unit: participants]
  Black or African American | 115
  White | 203
  Asian | 6
  American Indian/ Alaska Native | 2
  Other | 6
  Not Disclosed | 3
Region of Enrollment [Number; unit: participants]
  New Zealand | 9
  Canada | 26
  United States | 290
  Puerto Rico | 10
HCV Genotype [Number; unit: participants]
  Genotype 1a | 250
  Genotype 1b | 77
  Genotype 4 | 8
Cirrhosis Status [Number; unit: participants]
  No | 268
  Yes | 67
IL28b Status [Number; unit: participants] — The CC, CT, and TT alleles are different forms of the IL28b gene.
  participants
    CC | 81
    CT | 185
    TT | 69
Baseline HCV RNA [Mean (Standard Deviation); unit: log10 IU/mL] | 6.7 (0.64)
Baseline HCV RNA Category [Number; unit: participants]
  < 800,000 IU/mL | 36
  ≥ 800,000 IU/mL | 299
Baseline Serum Creatinine [Mean (Standard Deviation); unit: mg/dL] | 1.00 (0.210)
Estimated Glomerular Filtration Rate Using the Cockcroft-Gault Equation [Mean (Standard Deviation); unit: mL/min] | 101.6 (30.78)
Baseline CD4 Count [Mean (Standard Deviation); unit: cells/uL] | 662 (293.8)
Prior HCV Treatment [Number; unit: participants] — Acronyms for prior treatment:
  DAA = direct-acting antiviral; Peg-IFN = pegylated interferon; RBV = ribavirin
  participants
    Treatment-Naive | 150
    Treatment-Experienced with DAA+Peg-IFN+RBV | 53
    Treatment-Experienced with Peg-IFN+RBV | 113
    Treatment-Experienced with DAA+RBV | 14
    Treatment-Experienced with Other | 5

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Sustained Virologic Response (SVR) 12 Weeks After Discontinuation of Therapy (SVR12)
Description: SVR12 was defined as HCV RNA < the lower limit of quantitation (LLOQ; ie, 25 IU/mL) at 12 weeks after stopping study treatment.
Time Frame: Posttreatment Week 12
Population: Full Analysis Set: participants who enrolled and received at least 1 dose of study drug.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- LDV/SOF 12 Weeks: Primary Study: LDV/SOF (90/400 mg) FDC tablet once daily for up to 12 weeks.
Arm/Group | LDV/SOF 12 Weeks
Number analyzed (Participants) | 335
percentage of participants | 96.1 [93.5 to 97.9]

2. Primary Outcome: Percentage of Participants Who Permanently Discontinued Any Study Drug Due to an Adverse Event
Time Frame: Up to 12 weeks
Population: Safety Analysis Set: participants who enrolled and received at least 1 dose of study drug.
Measure: Number; unit: percentage of participants
Arm/Group | LDV/SOF 12 Weeks
Number analyzed (Participants) | 335
percentage of participants | 0

3. Secondary Outcome: Percentage of Participants With SVR at 4 and 24 Weeks After Discontinuation of Therapy (SVR4 and SVR24)
Description: SVR4 and SVR 24 were defined as HCV RNA < LLOQ at 4 and 24 weeks after stopping study treatment, respectively.
Time Frame: Posttreatment Weeks 4 and 24
Population: Full Analysis Set
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | LDV/SOF 12 Weeks
Number analyzed (Participants) | 335
percentage of participants
  SVR4 | 96.7 [94.2 to 98.3]
  SVR24 | 96.1 [93.5 to 97.9]

4. Secondary Outcome: Percentage of Participants With HCV RNA < LLOQ at Weeks 1, 2, 4, 6, 8, 10, and 12
Time Frame: Weeks 1, 2, 4, 6, 8, 10, and 12
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | LDV/SOF 12 Weeks
Number analyzed (Participants) | 335
percentage of participants
  Week 1 (N = 335) | 29.3 [24.4 to 34.4]
  Week 2 (N = 335) | 81.2 [76.6 to 85.2]
  Week 4 (N = 335) | 98.8 [97.0 to 99.7]
  Week 6 (N = 335) | 99.1 [97.4 to 99.8]
  Week 8 (N = 334) | 99.4 [97.9 to 99.9]
  Week 10 (N = 332) | 100.0 [98.9 to 100.0]
  Week 12 (N = 332) | 100.0 [98.9 to 100.0]

5. Secondary Outcome: Change From Baseline in HCV RNA at Weeks 1, 2, 4, 6, and 8
Time Frame: Baseline; Weeks 1, 2, 4, 6, and 8
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: log10 IU/mL
Arm/Group | LDV/SOF 12 Weeks
Number analyzed (Participants) | 335
log10 IU/mL
  Change at Week 1 (N = 331) | -4.68 (0.674)
  Change at Week 2 (N = 334) | -5.21 (0.654)
  Change at Week 4 (N = 335) | -5.30 (0.743)
  Change at Week 6 (N = 334) | -5.30 (0.772)
  Change at Week 8 (N = 333) | -5.33 (0.645)

6. Secondary Outcome: Percentage of Participants With Virologic Failure
Description: Virologic failure was defined as:
  * On-treatment virologic failure:
    * Breakthrough (confirmed HCV RNA ≥ LLOQ after having previously had HCV RNA < LLOQ while on treatment), or
    * Rebound (confirmed > 1 log10 IU/mL increase in HCV RNA from nadir while on treatment), or
    * Non-response (HCV RNA persistently ≥ LLOQ through 8 weeks of treatment)
  * Virologic relapse:
    * Confirmed HCV RNA ≥ LLOQ during the posttreatment period having achieved HCV RNA < LLOQ at last on-treatment visit.
Time Frame: Up to Posttreatment Week 24
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | LDV/SOF 12 Weeks
Number analyzed (Participants) | 335
percentage of participants
  On-Treatment Virologic Failure (N = 335) | 0.6
  Virologic Relapse (N = 333) | 3.0

7. Secondary Outcome: Percentage of Participants That Maintain HIV-1 RNA < 50 Copies/mL While on HCV Treatment
Time Frame: Weeks 4, 8, and 12
Population: Participants in the Safety Analysis Set with available data were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | LDV/SOF 12 Weeks
Number analyzed (Participants) | 335
percentage of participants
  Week 4 (N = 335) | 98.5
  Week 8 (N = 334) | 98.2
  Week 12 (N = 334) | 97.9

8. Secondary Outcome: Change From Baseline in Serum Creatinine at the End of Treatment (Week 12) and at Posttreatment Weeks 12 and 24
Time Frame: Baseline; Week 12, Posttreatment Weeks 12 and 24
Population: Participants in the Safety Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | LDV/SOF 12 Weeks
Number analyzed (Participants) | 335
mg/dL
  Change at Week 12 (N = 320) | 0.05 (0.111)
  Change at Posttreatment Week 12 (N = 325) | 0.03 (0.143)
  Change at Posttreatment Week 24 (N = 313) | -0.02 (0.134)

9. Secondary Outcome: For Participants in the Retreatment Substudy, Percentage of Participants With SVR at 4, 12, and 24 Weeks After Discontinuation of Therapy (SVR4, SVR12, and SVR24)
Description: SVR4, SVR12, and SVR 24 were defined as HCV RNA < LLOQ at 4, 12, and 24 weeks after stopping study treatment, respectively.
Time Frame: Posttreatment Weeks 4, 12, and 24 of Retreatment Substudy
Population: Participants in the Full Analysis Set who entered the Retreatment Substudy were analyzed.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- LDV/SOF+RBV 24 Weeks (Retreatment Substudy): Participants who experienced confirmed post-treatment virologic failure (relapse) at or before Posttreatment Week 24 during the Primary Study were eligible to be enrolled in the Retreatment Substudy to receive LDV/SOF (90/400 mg) FDC tablet once daily + RBV tablets (1000-1200 mg daily based on weight) for 24 weeks.
Arm/Group | LDV/SOF+RBV 24 Weeks (Retreatment Substudy)
Number analyzed (Participants) | 9
percentage of participants
  SVR4 | 88.9 [51.8 to 99.7]
  SVR12 | 88.9 [51.8 to 99.7]
  SVR24 | 88.9 [51.8 to 99.7]

10. Secondary Outcome: For Participants in the Retreatment Substudy, Percentage of Participants With HCV RNA < LLOQ at Retreatment Weeks 2, 4, 8, 12, 16, 20, and 24
Time Frame: Weeks 2, 4, 8, 12, 16, 20, and 24 of the Retreatment Substudy
Population: Participants in the Full Analysis Set who entered the Retreatment Substudy were analyzed.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | LDV/SOF+RBV 24 Weeks (Retreatment Substudy)
Number analyzed (Participants) | 9
percentage of participants
  Week 2 Retreatment | 88.9 [51.8 to 99.7]
  Week 4 Retreatment | 100.0 [66.4 to 100.0]
  Week 8 Retreatment | 100.0 [66.4 to 100.0]
  Week 12 Retreatment | 100.0 [66.4 to 100.0]
  Week 16 Retreatment | 100.0 [66.4 to 100.0]
  Week 20 Retreatment | 100.0 [66.4 to 100.0]
  Week 24 Retreatment | 100.0 [66.4 to 100.0]

11. Secondary Outcome: For Participants in the Retreatment Substudy, Change From Baseline in HCV RNA at Retreatment Weeks 2, 4, and 8
Time Frame: Baseline; Weeks 2, 4, and 8 of Retreatment Substudy
Population: Participants in the Full Analysis Set who entered the Retreatment Substudy were analyzed.
Measure: Mean (Standard Deviation); unit: log10 IU/mL
Arm/Group | LDV/SOF+RBV 24 Weeks (Retreatment Substudy)
Number analyzed (Participants) | 9
log10 IU/mL
  Change at Week 2 Retreatment | -5.01 (0.775)
  Change at Week 4 Retreatment | -5.04 (0.802)
  Change at Week 8 Retreatment | -5.04 (0.802)

12. Secondary Outcome: For Participants in the Retreatment Substudy, Percentage of Participants With Virologic Failure
Description: as for outcome 6
Time Frame: Up to Posttreatment Week 24 of Retreatment Substudy
Population: Participants in the Full Analysis Set who entered the Retreatment Substudy were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | LDV/SOF+RBV 24 Weeks (Retreatment Substudy)
Number analyzed (Participants) | 9
percentage of participants
  On-Treatment Virologic Failure | 0
  Virologic Relapse | 11.1

ADVERSE EVENTS:
Time Frame: LDV/SOF 12 Weeks: Up to 12 weeks plus 30 days; LDV/SOF+RBV 24 Weeks: Up to 24 weeks plus 30 days
Description: Safety Analysis Set
Groups:
- LDV/SOF 12 Weeks (Primary Study): LDV/SOF (90/400 mg) FDC tablet once daily for up to 12 weeks.
- LDV/SOF+RBV 24 Weeks (Retreatment): Participants who experienced confirmed post-treatment virologic failure (relapse) at or before Posttreatment Week 24 during the Primary Study were eligible to be enrolled in the Retreatment Substudy to receive LDV/SOF (90/400 mg) FDC tablet once daily + RBV tablets (1000-1200 mg daily based on weight) for 24 weeks.
Arm/Group | LDV/SOF 12 Weeks (Primary Study) | LDV/SOF+RBV 24 Weeks (Retreatment)
Serious Adverse Events (participants affected / at risk) | 8/335 | 0/9
Other Adverse Events (participants affected / at risk) | 179/335 | 9/9
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | LDV/SOF 12 Weeks (Primary Study) (N=335) | LDV/SOF+RBV 24 Weeks (Retreatment) (N=9)
Diarrhoea (Gastrointestinal disorders) | 1 | 0
Ileus (Gastrointestinal disorders) | 1 | 0
Portal vein thrombosis (Hepatobiliary disorders) | 2 | 0
Clostridium difficile colitis (Infections and infestations) | 1 | 0
Peritonitis bacterial (Infections and infestations) | 1 | 0
Respiratory tract infection (Infections and infestations) | 1 | 0
Sepsis (Infections and infestations) | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Hepatocellular carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Substance abuse (Psychiatric disorders) | 1 | 0
Azotaemia (Renal and urinary disorders) | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | LDV/SOF 12 Weeks (Primary Study) (N=335) | LDV/SOF+RBV 24 Weeks (Retreatment) (N=9)
Anaemia (Blood and lymphatic system disorders) | 2 | 3
Haemolytic anaemia (Blood and lymphatic system disorders) | 0 | 1
Vision blurred (Eye disorders) | 2 | 1
Diarrhoea (Gastrointestinal disorders) | 35 | 1
Nausea (Gastrointestinal disorders) | 33 | 1
Vomiting (Gastrointestinal disorders) | 14 | 1
Fatigue (General disorders) | 71 | 6
Chest discomfort (General disorders) | 0 | 1
Cyst (General disorders) | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 18 | 1
Acute sinusitis (Infections and infestations) | 0 | 1
Blood uric acid increased (Investigations) | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 8 | 1
Increased appetite (Metabolism and nutrition disorders) | 1 | 1
Abnormal loss of weight (Metabolism and nutrition disorders) | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 23 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 7 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 3 | 1
Foot deformity (Musculoskeletal and connective tissue disorders) | 0 | 1
Headache (Nervous system disorders) | 82 | 1
Dizziness (Nervous system disorders) | 11 | 1
Irritability (Psychiatric disorders) | 10 | 1
Emotional disorder (Psychiatric disorders) | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 8 | 4
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Nasal dryness (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 4 | 1
Dry skin (Skin and subcutaneous tissue disorders) | 2 | 1
Ingrowing nail (Skin and subcutaneous tissue disorders) | 1 | 1
Rash generalised (Skin and subcutaneous tissue disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
After conclusion of the study and without prior written approval from Gilead, investigators in this study may communicate, orally present, or publish in scientific journals or other media only after the following conditions have been met:

* The results of the study in their entirety have been publicly disclosed by or with the consent of Gilead in an abstract, manuscript, or presentation form; or
* The study has been completed at all study sites for at least 2 years